CLINICAL TRIAL: NCT06435338
Title: Patient Decision Aid Tool for HPV Vaccination Among Adults Ages 27-45 Years Old
Acronym: HPV Decide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: University of North Texas Health Science Center (Other); University of South Florida (Other); Temple University (Other); Indiana University School of Medicine (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Erika L. Thompson, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 100257
Record Dates: First submitted 2024-05-20; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Decision Aid; Hpv
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient decision aid (Experimental): Patient decision aid on HPV vaccination on webpage.
  Interventions: Behavioral: Patient decision aid
- Control (Active Comparator): Vaccine information sheet on HPV vaccination view on webpage.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Patient decision aid — The patient decision aid for HPV vaccination among mid-adults, named HPV Decide. It is delivered online on a website.
  Arms: Patient decision aid
Behavioral: Control — Vaccine information sheet on HPV vaccination. Attention control condition.
  Arms: Control

SUMMARY:
The goal of this study is to learn if a patient decision tool for HPV vaccination works for decision-making among adults ages 27-45. Researchers will compare a web-based patient decision tool to an information sheet to see if the tool works for decision-making. Participants will take a baseline survey, view the intervention or control condition, and then take a follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

* Unvaccinated for HPV
* 27-45 years
* Resides in the United States
* Reads English
* Consents to participate

Exclusion Criteria:

* none

Ages: 27 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cis-gender male or female only due to randomization stratification
Enrollment: 632 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Decisional conflict - 16 item scale | Immediate post-test
  This scale has 16 items and 5 response categories. The decisional conflict scale (DCS) measures personal perceptions of: uncertainty in choosing options; modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making; and effective decision making (in full version) such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice. The scores ranged from 0 "no conflict" to 100 "extreme decisional conflict."
Decisional conflict - 4 item scale | Immediate post-test
  Decision conflict scale recommended for every day clinical practice. It has 4 items and two response categories. Scores range from 0 [extremely high decisional conflict] to 4 [no decisional conflict].

SECONDARY OUTCOMES:
Knowledge | Immediate post-test
  16-item knowledge item related to human papillomavirus and human papillomavirus vaccination. Scale from 0 [low knowledge] to 16 [high knowledge].
Intentions | Immediate post-test
  Intentions for information seeking, talking to a healthcare provider, and getting vaccinated
Decision | Immediate post-test
  Vaccine decision, including decide to get vaccinated, unsure, and decided not to get vaccinated
Perceived expectation | Immediate post-test
  Perceived expectation was assessed by asking participant agreement on a 5-point Likert scale to the following statement, "The effectiveness of the HPV vaccine will vary from person to person." Higher score indicates higher perceived effectiveness.
Perceived risk | Immediate post-test
  Perceived risks of HPV infection were also assessed, including participants' perceptions of getting an HPV-associated infection genital/anal warts, or cancer in their lifetime. Response options ranged from very unlikely (lower score) to very likely (higher score).
  How likely are you to get an HPV related cancer, like cervical, oral, or anal cancer, in your lifetime? How likely are you to get an HPV infection in your lifetime? How likely are you to get anal or genital warts in your lifetime?
Decision self-efficacy | Immediate post-test
  The Decision Self-Efficacy Scale evaluates an individual's self-confidence to make decisions on their own or with support from other sources. Scores range from 0 [extremely low self-efficacy] to 100 [extremely high self efficacy].

CONTACTS AND LOCATIONS:
Locations (1):
- UT School of Public Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request to the PI, study materials will be shared.

REFERENCES:
- [Background] O'Connor AM. User Manual - Decisional Conflict Scale (16 item question format). Ottawa: Ottawa Hospital Research Institute. 1993. http://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Decisional_Conflict.pdf
- [Background] Legare F, Kearing S, Clay K, Gagnon S, D'Amours D, Rousseau M, O'Connor A. Are you SURE?: Assessing patient decisional conflict with a 4-item screening test. Can Fam Physician. 2010 Aug;56(8):e308-14. PMID 20705870
- [Background] O'Connor AM. User Manual - Decision Self-Efficacy Scale. Ottawa: Ottawa Hospital Research Institute. 1993. http://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Decision_SelfEfficacy.pdf
- [Background] Garg A, Wheldon CW, Galvin AM, Moore JD, Griner SB, Thompson EL. The Development and Psychometric Evaluation of the Mid-adult Human Papillomavirus Vaccine Knowledge Scale in the United States. Sex Transm Dis. 2022 Jun 1;49(6):423-428. doi: 10.1097/OLQ.0000000000001615. Epub 2022 Feb 8. PMID 35608097
- [Derived] Thompson EL, Luningham J, Alkhatib SA, Grace J, Akpan IN, Daley EM, Zimet GD, Wheldon CW. Testing an HPV Vaccine Decision Aid for 27- to 45-Year-Old Adults in the United States: A Randomized Trial. Med Decis Making. 2025 Feb;45(2):192-204. doi: 10.1177/0272989X241305142. Epub 2024 Dec 24. PMID 39717960